CLINICAL TRIAL: NCT05386446
Title: Prospective Open Controlled Non-interventional Study of the Use of the Drug Ingaron (Interferon Gamma Human Recombinant, NPP Farmaklon LLC, Russia) in Volunteers for the Prevention of Coronavirus Infection COVID-19
Brief Title: Study of the Use of the Ingaron in Volunteers for the Prevention of COVID-19
Status: Completed | Type: Observational
Sponsor: SPP Pharmaclon Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: GAMMACOVID-PROF
Record Dates: First submitted 2022-05-20; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Respiratory Infection
Keywords: COVID-19 prevention; interferon gamma; nasal drops

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drug: Interferon Gamma: Ingaron (INN: recombinant human interferon gamma, lyophilisate for solution for intranasal administration 100,000 IU) in the regime of 3 drops in each nasal passage intranasally every other day for 10 days with a break of 7 days (2 10-day cycles)
  Interventions: Drug: Interferon gamma human recombinant (IFN-G)
- Control: No intervention: Любой профилактический метод, включающий различные фармакологические методы лечения COVID-19, наряду с применением противовирусных и иммуномодулирующих средств, за исключением препаратов, назначаемых не по назначению или в исследовательских целях, а также IFN-G.

INTERVENTIONS:
Drug: Interferon gamma human recombinant (IFN-G) — nasal form
  Other Names: Ingaron; Interferon gamma human recombinant
  Groups: Drug: Interferon Gamma

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of the prophylactic use of Ingaron (INN: recombinant interferon gamma human, lyophilisate for solution for intranasal administration 100,000 IU) in the regimen of 3 drops in each nasal passage intranasally every other day for 10 days with a break of 7 days (2 10-day cycles) in volunteers.

DETAILED DESCRIPTION:
Distribution between groups is made randomly at the request of the participant. According to the methodology approved by the observational program, the participant must use or not use the investigational drug (depending on the distribution group and their own will) during the 27 days of the prophylaxis course (10 days + 7 days + 10 days). The control group does not receive study therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Medical workers and medical personnel working in the "red zone" and in contact with patients infected with COVID-19.
2. Men and women over 18 years of age.
3. Signing an informed consent form for data processing.
4. Ability and agreement to complete the questionnaire (part 1) of the participant.
5. No symptoms of a respiratory infection.
6. Negative PCR test result for the presence of SARS-CoV-2 RNA according to the biomaterial obtained by nasopharyngeal swab.

Exclusion Criteria:

1. Any clinically confirmed or documented history of diseases that may complicate the interpretation of the data being assessed (HIV, cancer, organ transplantation, etc.).
2. Any other comorbidities or conditions that, in the opinion of the investigator, may distort the results of the study, limit the rights of the volunteer, or put him at greater risk.
3. Contraindications to the use of the investigational medicinal product.
4. Individual intolerance to the ingredients that make up the study drug.
5. Pregnancy or breastfeeding.
6. The presence of antibodies to SARS-CoV-2 (IgM, IgG).

Ages: 21 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Volunteers working in the "red zone" with patients infected with SARS-CoV-2
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence rate | Day 35
  The incidence rate of COVID-19 volunteers when using the drug Ingaron (INN: interferon gamma human recombinant, lyophilisate for solution for intranasal administration 100,000 IU) in the regimen of 3 drops in each nasal passage intranasally every other day for 10 days with a break of 7 days ( 2 10-day cycles) vs control group

SECONDARY OUTCOMES:
Frequency of laboratory confirmation of COVID-19 disease | Day 35
  The frequency of laboratory confirmations of COVID-19 disease when using Ingaron (INN: recombinant human interferon gamma, lyophilisate for solution for intranasal administration 100,000 IU) in the regimen of 3 drops in each nasal passage intranasally every other day for 10 days with a break of 7 days (2 10-day cycles) vs control group
Comparative assessment of scores on the WHO scale (0-8) | Day 35
  Comparative evaluation of scores on the WHO scale (from 0 points - not infected, no manifestations or virological signs of infection, up to 8 points - died, death) when using the drug Ingaron (INN: interferon gamma human recombinant, lyophilisate for solution for intranasal administration 100,000 IU) in the mode of 3 drops in each nasal passage intranasally every other day for 10 days with a break of 7 days (2 10-day cycles) in comparison with the control group
Severity of symptoms | Day 35
  The severity of symptoms of the disease of infected study participants in both groups
Duration of symptoms | Day 35
  The duration of symptoms of the disease of infected study participants in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly I Saulin, Master, Study Director — SPP Pharmaclon Ltd.
Locations (1):
- City Clinical Hospital named after M.E. Zhadkevich Moscow City Health Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myasnikov AL, Berns SA, Zverev KV, Lartseva OA, Talyzin PA. Efficacy of Interferon Gamma in the Prevention of SARS-CoV-2 Infection (COVID-19): Results of a Prospective Controlled Trial. International Journal of Biomedicine 2020; 10(3): 182-188.